CLINICAL TRIAL: NCT07350239
Title: Prospective Clinical, Microbial and Tissue-based Characterization Analyses of Severe Temporomandibular Joint Pathology
Brief Title: Clinical, Microbial and Tissue-based Characterization of Patients Treated for Severe Temporomandibular Joint Pathology
Status: Not yet recruiting | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00596-01
Record Dates: First submitted 2025-01-07; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: TMJ Disorder; Ankylosis; Osteoarthritis
Keywords: TMJ; Temporomandibular joint; TMJ disorder; oral and maxillafacial surgery; TMJ pain; TMJ ankylosis; Severe osteoarthritis
MeSH Terms: conditions — Temporomandibular Joint Disorders; Ankylosis; Osteoarthritis; Temporomandibular ankylosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbial DNA analysis will be executed on both soft tissue samples and fresh frozen bone tissue. (16S rRNA Sequencing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with TMJ ankylosis or severe osteoarthritis of TMJ.
  Interventions: Procedure: open TMJ surgery such as arthroplasty surgery with or without autogen or allogen reconstruction

INTERVENTIONS:
Procedure: open TMJ surgery such as arthroplasty surgery with or without autogen or allogen reconstruction — Consecutive patients (n=20) were offered open TMJ surgery, such as arthroplasty surgery with or without autogenous or allogenic reconstruction, due to TMJ ankylosis or severe osteoarthritis. The patients were treated at Karolinska University Hospital, Örebro University Hospital, or Lund University Hospital.

SUMMARY:
The general objective of this observational study is to clarify the clinical, microbial, and tissue characteristics, aetiology, and risk factors behind severe TMJ pathology. The main questions it aims to answer are:

* What are the clinical and histologic characteristics of patients with severe pathology of the TMJ?
* Can microbial DNA be found in TMJ tissue from patients with severe pathology of the TMJ, and if so, does this correlate to the outcome of the surgery?

DETAILED DESCRIPTION:
The temporomandibular joint (TMJ) is a synovial joint characterized by a combination of rotation and translation during mouth opening. Unlike other joints in the body, the joint cartilage is fibrous and innervated by cranial nerves. Normal TMJ function is essential for vital functions such as eating, including proper mouth opening capacity, as well as for social activities such as talking, laughing, singing, and kissing. Several studies have reported a severe impact on the quality of life for patients with impaired and painful TMJ function.

Temporomandibular joint disorders (TMD) are common, affecting approximately 20% of the population with a strong, as yet unexplained, female predominance. The aetiology of internal derangement of the TMJ is unknown, but trauma and local or general joint hypermobility have been discussed as possible predisposing factors.

In a small proportion of patients, severe TMJ pathology, including ankylosis, develops. If ankylosis occurs, the condylar process of the mandible becomes fused to the fossa by fibrotic or bony tissue, resulting in severely restricted mouth opening ability. This can lead to a total inability to move the jaw, which can, in turn, be potentially life-threatening due to compromised airways in case of nausea.

In developing countries, TMJ ankylosis usually develops during early childhood as a complication of otitis media (inflammation of the middle ear). In the industrialized world, the condition is more frequent in adults. Factors suggested to cause severe TMJ disease, including ankylosis, are local or systemic infections or rheumatic diseases. According to some studies, a common etiological factor is trauma through intra-articular hematoma, tissue scarring, and excessive bone formation. Since most TMJ trauma resolves uneventfully, this does not explain the individual susceptibility to developing severe TMJ pathology. Thus, the aetiology and epidemiology of these conditions remain unknown.

Previous data point in different directions regarding the role of bacteria in TMJ pathology. However, knowledge regarding the role of chronic, low-virulent microbial challenges in post-surgically deteriorating cases with severe arthritis or ankylosis is lacking. Furthermore, the histopathologic presentation of these conditions is largely unknown, and systematic approaches for tissue categorization and diagnostics are lacking.

There are different surgical procedures available for these severe TMJ conditions, including osteoarthrectomy (removal of the joint bone), interpositional osteoarthrectomy using the temporalis muscle, and/or joint reconstruction using alloplastic materials or autogenous grafts. The choice of surgical technique is debated, and supporting long-term follow-up studies are lacking.

Previous studies have mainly focused on surgical interventions in a series of patients with TMJ disease without accounting for diagnosis or clinical presentation, leading to uncertainties regarding treatment decisions and efficacy. Knowledge of the mechanisms behind severe TMJ disease will improve the understanding, prediction, management, and prognosis of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to open TMJ surgery such as arthroplastic surgery with or without autogen or allogen reconstruction
* Preserved biobank material (resected bone and soft tissue).

Exclusion Criteria:

* Absence of biobank material.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients (n=20) offered open TMJ surgery such as arthroplasty surgery with or without autogen or allogen reconstruction due to TMJ ankyloses or severe osteoarthritis. Patients treated at Karolinska University Hospital, Örebro University Hospital or Lund University Hospital. Exclusion criteria: suspicion of malignancy, inability to give consent.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical investigation (patients): | Inclusion will take at least 3 years, followed by one year of follow-up
  Preoperatively, 1 week postoperatively, and at 1, 3, 6, and 12 months, or at the last visit after surgery, objective measures according to clinical routines for TMJ internal derangement patients will be collected. MRI and/or CBCT/CT will be performed preoperatively. Subjective measures include scoring functional severity and grading symptoms according to a 10-point visual analogue scale (VAS) in terms of pain intensity, functional disability, and psychosocial impact.
Questionnaires: | Inclusion will take at least 3 years, followed by one year of follow-up.
  Three questionnaires: Oral Health Impact Profile-14 (OHIP-14), Jaw Function Limitation Scale-8 (JFLS-8), and EuroQol-5D-5L will be distributed to the patients. The patients will complete the questionnaires at the first visit and at the one-year follow-up after surgery. All three questionnaires are validated and available in Swedish.
  OHIP-14: 14 questions answered on the scale:
  - Does not apply to me, Very often, Quite often, Sometimes, Rarely, Never.
  JFLS-8: 8 questions answered on the scale:
  - 0 (no limitation) up to 10 (major limitation).
  EuroQol-5D-5L: 5 questions, each with 5 options, that can be answered with:
  - Yes or No."
Histopathologic analyses: | 3 years
  Fresh specimens from resected TMJ tissue will be processed with formalin fixation (4%) for a minimum of 48 hours and sent to the Pathology department. The tissue will be decalcified with 7% formic acid for 2-4 weeks. The decision to arrest the decalcification process will depend on the softness of the tissue, which will be assessed by using the ability of a needle to transpierce the sample. Thereafter, the specimens will be dehydrated and paraffin-embedded according to routine procedures. For routine histological diagnoses, 3 μm thick sections will be stained with hematoxylin and eosin. Immunohistochemistry staining, as well as other complementary staining methods, will be performed using antibodies based on the results of the retrospective analyses. Part of the specimens will be fresh frozen.
  A specialist in pathology will review all the samples, categorize them, and assess them to identify any common denominators between the samples.
Analysis of microbial DNA in the Biobank material using 16S metagenomic sequencing | 3 years
  Microbial DNA analyses will be performed on formalin-fixed paraffin-embedded (FFPE) soft tissue specimens from the biobank. DNA will be purified using the QIAamp DNA FFPE Advanced UNG Kit (Qiagen) with an additional bead-beating step. The full-length 16S rRNA gene (variable V1-V9 regions) will be sequenced to identify the bacterial organisms at the species level. Amplification of the 16S rRNA gene (~1500bp) and library preparation will be performed using the 16S Barcoding Kit (Oxford Nanopore Technology, ONT), allowing multiplexing of samples and thereby reducing costs.
  Specialists in molecular biology and bioinformaticians will handle the results. Everything, from whether bacterial DNA is found to which different bacteria are present in what quantities, will be noted.
Objective & Subjective measurements | Inclusion will take at least 3 years. Then one year follow up
  Registration:
  (Specify in writing)
  * Past and current diseases
  * Medication
  * Medicational allergy
  Preoperative information registered at the initial visit:
  * TMJ trauma (yes/no)
  * TMJ dislocation (yes/no)
  * Parafunction (None/ Grinding/ Clenching)
  Preoperative Symptoms (Initial Visit, Subjective)
  * Crepitation: (Right/Left)
  * Clicking/Locking: (Right/Left)
  * Locking: (Right/Left)
  * Movement Pain: (Right/Left)
  * Restricted Mouth Opening: (Right/Left)
  * Difficulty Eating: (yes/no)
  * Difficulty Speaking: (yes/no)
  * Other: (write in text)
  Preoperative TMJ-Related Treatment
  * None
  * Conservative treatment: Bite splint, movement training, NSAIDs, bite correction, occlusal therapy
  * Corticosteroid injection
  * Arthrocentesis
  * Arthroscopy: Date (year & which joint):
  * Open joint surgery: (If previous surgery, specify which and year)
  * Other treatments
  Surgery:
  * Surgical date
  * Age at surgery
  * Type of surgery
  * Surgical side (Right/left/bilateral)
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  The following measures will be recorded using the Visual Analog Scale (VAS) of 0-10:
  TMJ Pain During Function:
  * Measured on a scale from 0 to 10 for pain intensity.
  * Right/left TMJ will be assessed separately.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  Palpation Tenderness Over the Temporomandibular Joints Laterally:
  * Scale: Yes/No for tenderness.
  * Right/Left TMJ.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
  Palpation Tenderness Over the Masticatory Muscles (Pain Rating >2 on the Same Side):
  * Scale: Yes/No for tenderness.
  * Right/Left TMJ.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  The following measures will be recorded using the Visual Analog Scale (VAS) of 0-10:
  Functional Impairment (Eating, Chewing, Biting)
  * Measured on a scale from 0 to 10 for difficulty in performing these functions.
  * Right/left TMJ will be assessed separately.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  The following measures will be recorded using the Visual Analog Scale (VAS) of 0-10:
  Global Pain:
  * Measured on a scale from 0 to 10 for overall pain experience.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  The following measures will be recorded using the Visual Analog Scale (VAS) of 0-10:
  Psycho-social Influence:
  * Measured on a scale from 0 to 10 for the psychological or social impact of pain and dysfunction.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  Maximal Interincisal Opening:
  * Scale: Measured in millimeters.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
  Maximal Lateral Movement (TMJ):
  * Measured in millimeters.
  * Right/Left TMJ.
  * Time points: Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.

SECONDARY OUTCOMES:
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  Occlusal Relationships:
  * Written description of the occlusal relationship.
  * Time points: Preoperative and 1 year postoperative
Objective and subjective measurments | Inclusion will take at least 3 years. Then one year follow up
  Postoperative Complications
  * Written description of complications:
  * Nerve Damage: Yes/No, and specify if transient (with duration) or permanent.
  * Infection: Yes/No, and specify treatment (if any).